CLINICAL TRIAL: NCT04536779
Title: "When Movement Moves" - A Self-controlled Trial of the Physiological, Mental and Social Health Benefits Among Individuals With Low Physical Mobility Moved by Others in Two Existing Initiatives: the Danish Team Twin and Cycling Without Age
Brief Title: "When Movement Moves" - The Health Benefits Among Individuals With Low Physical Mobility Moved by Others
Acronym: WMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Rigshospitalet, Denmark (Other); Bevica Fonden (Other); Sygekassernes Helsefond (Other)
Responsible Party: Principal Investigator, Christina Bjørk Petersen, Associate Professor, University of Southern Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19/66334
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Physical Disability; Healthy
Keywords: non-elite sports community; physically challenged; individuals with low physical mobility; volunteers; relatives; disabled; QOL

STUDY DESIGN:
Intervention Model Description: We will use a study design with pre- and post-measurements. The participant will be their own case-control. For optimizing the statistical strength, the individuals with low mobility will undergo two times of baseline measurements. After a minimum of a three-month trial period followup measurements will be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individuals with low mobility (Disabled and Elder) (Experimental): minimum 8-10 training sessions in at least three months.
  Interventions: Other: Training in the local departments of TT and cycling trips with CUA

INTERVENTIONS:
Other: Training in the local departments of TT and cycling trips with CUA — in a minimum of 3 months, the individuals with low physical mobility will conduct a minimum of 8-10 training and cycling sessions.

SUMMARY:
The purpose of the trial is to investigate the physiological, mental, social health effect among individuals with low physical mobility participating in one of the two pre-existing initiatives: the Danish 'Team Twin' and Cycling Without Age. In these, the individuals with low physical mobility are moved by and together with by normal functioning volunteers.

Based on the above, this research project will answer the following research questions:

1. Does movement by others improves the quality of life (QOL) among individuals with low physical mobility
2. Does movement by others improves the physiological health among individuals with low physical mobility
3. Does moving individuals with low physical mobility improve health among normal functioning individuals (i.e volunteer runners and pilots)?
4. How does participation in the physical activity initiatives influence well-being, relations and attitudes among relatives (to the disabled individuals) and employees at nursing homes?

DETAILED DESCRIPTION:
The research project consists of two sub-projects, where data collection will take place independently of each other. For both projects, we will use a self-controlled study design with pre- and post-measurements of the participant. Through a mixed-method design combining both quantitative and qualitative data will be obtained from the following three target groups:

1. Individuals with low physical mobility (referred to as 'Handiathletes' in the TT-subproject and 'Passengers' in the CUA-sub project)
2. Volunteers (Runners and Pilots)
3. Relatives (to the Handiathletes) and employees at nursing homes (older people)

I collaboration with the two initiatives: the Team Twin- & Cycling without Age-foundation, the study intend to recruit approximately 25 'Handiathletes' and 25 'Passengers' with low physical mobility and a non-defined number of volunteer-runners, pilots and relatives from most recent established local departments of TT and nursing homes who offers the CUA-concepts to the nursing home residents. Prior to the enrollment, all participants will be given oral and written participant information and give their written consent to participate. Depending on the target group, each group will undergo different data collection methods (described under outcome).

Team Twin description:

Primo 2021, the Handiathletes (TT) who meet eligibility criteria will undergo two clinical pre-test days within a two weeks interval. Starting from approximately ultimo February, a training period of minimum 3 months will start. All the participant target groups train and participate in prescheduled races in their respective departments of TT. During the 3 months of training, data will be collected from the different target groups (see outcome measure). After the 3 months of training, the 'Handiathletes' will undergo one clinical post-test.

The Cycling Without Age description:

Primo 2021, the Pilots (CUA) who meet eligibility criteria will be enrolled in the project - a trial period of minimum 3 months. We will conduct pre- and post measures regarding the research questions (described under outcome)

ELIGIBILITY:
Inclusion Criteria:

Disabled from the departments of TT:

- Pass the medical examination conducted by the responsible investigator at the laboratory.

Volunteers;

* Active member of a local department of TT
* Volunteer in Cycling without Age

Relatives and nursing home employees;

* Relative to the enrolled disabled participant
* working at a nursing home who offers CUA

Exclusion Criteria:

- Sustain damage, which makes the person unable to continue the training sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Quality Of Life (QOL) | Baseline to follow-up
  Validated self-reported measure of quality of life (i.e. Cantril Ladder)

SECONDARY OUTCOMES:
Physiological Health | Baseline to follow-up
  Measured objectively and by self-report:
  * Cardiorespiratory and metabolic fitness
  * Cognitive and physical functioning
  * Quantity and severity of symptoms related to their disease/disability
  * Sleep quality and duration
Mental Health | Baseline to follow-up
  Measured by self-reported questionnaire and interviews:
  * wellbeing and life satisfaction
  * loneliness
  * Acceptance and coping (learn to live with diagnosis)
Social Health | Baseline to follow-up
  Measured by interviews and self-reported questionnaire:
  * Network, relations and Sense of Coherence (SOC)
  * Acceptance from surroundings
Autonomy | Baseline to follow-up
  Measured by interviews and self-reported questionnaire:
  * Independence in activities of daily living
  * Feeling of being in control of and taking act in one's own life
  * options and choices

CONTACTS AND LOCATIONS:
Overall Officials: Christina B Petersen, Assoc. Prof, Principal Investigator — National Institute of Public Health, SDU; Mette Toftager, Researcher, Principal Investigator — National Institute of Public Health, SDU
Locations (1):
- National institute of Public Health, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorgensen A, Petersen CB, Eghoj M, Toftager M. When Movement Moves: Study Protocol for a Multi-Method Pre/Post Evaluation Study of Two Programmes; the Danish Team Twin and Cycling Without Age. Int J Environ Res Public Health. 2021 Sep 23;18(19):10008. doi: 10.3390/ijerph181910008. PMID 34639309
- [Derived] Jorgensen A, Toftager M, Eghoj M, Ried-Larsen M, Bjork Petersen C. Heart rate responses, agreement and accuracy among persons with severe disabilities participating in the indirect movement program: Team Twin-an observational study. Front Sports Act Living. 2023 Oct 24;5:1213655. doi: 10.3389/fspor.2023.1213655. eCollection 2023. PMID 37941848
- See also: The Team Twin Foundation — https://teamtvilling.dk/
- See also: Cycling Without Age — https://cyklingudenalder.dk/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT04536779/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-13): https://cdn.clinicaltrials.gov/large-docs/79/NCT04536779/ICF_001.pdf